CLINICAL TRIAL: NCT00683202
Title: The Significance of Low-Dose Aspirin on Ovarian Responsiveness, Uterine Hemodynamics and Pregnancy Outcome in in Vitro Fertilization and in Intracytoplasmic Sperm Injection: A Randomized, Placebo-Controlled Double-Blind Study
Brief Title: Low-Dose Aspirin in in Vitro Fertilization (IVF) and Intracytoplasmic Sperm Injection (ICSI) Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Bayer (Industry); Kuopio University Hospital (Other); Tampere University (Other)
Responsible Party: Mervi Haapsamo/MD, University Hospital of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 56/2001
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2001-03

CONDITIONS: Pregnancy; Miscarriage Less Than 12 Gestational Weeks; Extrauterine Pregnancy; Preeclampsia; Intrauterine Fetal Growth Restriction
Keywords: Assisted reproduction; Ovarian response; Uteroplacental hemodynamics; Doppler ultrasonography; Implantation rate; Pregnancy rate; Live birth rate
MeSH Terms: conditions — Pregnancy, Ectopic; Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Acetylsalicylic acid 100 mg daily perorally
  Interventions: Drug: Acetylsalicylic acid
- 2 (Placebo Comparator): Placebo daily perorally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid — Acetylsalicylic acid 100 mg or placebo daily perorally started on the first day of ovarian gonadotrophin stimulation in in vitro fertilization or in intracytoplasmic sperm injection
  Other Names: Low-dose aspirin
  Arms: 1
Drug: Placebo — Acetylsalicylic acid 100 mg or placebo daily perorally started on the first day of ovarian gonadotrophin stimulation in in vitro fertilization or in intracytoplasmic sperm injection
  Arms: 2

SUMMARY:
In this study we hypothesized that low-dose aspirin therapy (100 mg daily) improves ovarian responsiveness, uterine haemodynamics and clinical pregnancy rates in unselected subjects undergoing IVF/ICSI when the treatment is started concomitantly with controlled ovarian hyperstimulation.

DETAILED DESCRIPTION:
Low-dose acetylsalicylic acid irreversibly inhibits the cyclo-oxygenase enzyme in platelets, thus preventing the synthesis of thromboxane, which causes vasoconstriction and platelet aggregation. By this mechanism low-dose aspirin may enhance ovarian and uterine blood flow and tissue perfusion and thus improve ovarian responsiveness for gonadotrophins and endometrial receptivity for implantation. Randomized controlled studies and meta-analyses on the low-dose aspirin therapy to improve IVF/ICSI outcome or uterine hemodynamics have revealed conflicting results.

ELIGIBILITY:
Inclusion Criteria:

* age < 40 years
* < 4 previous ovarian stimulations

Exclusion Criteria:

* allergy for acetylsalicylic acid

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2001-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | Five weeks after embryo transfer

SECONDARY OUTCOMES:
Uterine artery and spiral artery pulsatility index values | On the day of embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Mervi Haapsamo, MD, Principal Investigator — University Hospital of Oulu, Finland; Juha Rasanen, MD, Study Director — University Hospital of Oulu, Finland and Oregon Health Sciences University, Oregon USA; Hannu Martikainen, MD, Study Director — University Hospital of Oulu, Finland; Juha S Tapanainen, Prof, Study Director — University Hospital of Oulu, Finland; Seppo Heinonen, Prof, Study Director — University Hospital of Kuopio, Finland; Helena Tinkanen, MD, Study Director — Unversity Hospital of Tampere, Finland
Locations (1):
- University Hospital of Oulu, Department of Obstetrics and Gynecology, Oulu, Finland

REFERENCES:
- [Derived] Haapsamo M, Martikainen H, Tinkanen H, Heinonen S, Nuojua-Huttunen S, Rasanen J. Low-dose aspirin therapy and hypertensive pregnancy complications in unselected IVF and ICSI patients: a randomized, placebo-controlled, double-blind study. Hum Reprod. 2010 Dec;25(12):2972-7. doi: 10.1093/humrep/deq286. Epub 2010 Oct 13. PMID 20943705
- [Derived] Haapsamo M, Martikainen H, Rasanen J. Low-dose aspirin and uterine haemodynamics on the day of embryo transfer in women undergoing IVF/ICSI: a randomized, placebo-controlled, double-blind study. Hum Reprod. 2009 Apr;24(4):861-6. doi: 10.1093/humrep/den489. Epub 2009 Jan 18. PMID 19153091